CLINICAL TRIAL: NCT01116791
Title: Cytoreductive Surgery Plus Hyperthermic Intraoperative Peritoneal Chemotherapy With Cisplatin to Treat Peritoneal Carcinomatosis From Upper Gastrointestinal Cancer; the HIPCUpp-trial
Brief Title: Cytoreductive Surgery(CRS) Plus Hyperthermic Intraoperative Peritoneal Chemotherapy(HIPC) With Cisplatin to Treat Peritoneal Carcinomatosis From Upper Gastrointestinal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient enrollment in Pancreatic & Biliary arm
Sponsor: Baki Topal (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor-Investigator, Baki Topal, Professor of Surgery, University Hospital, Gasthuisberg
Organization: University Hospital, Gasthuisberg (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIPCUpp-trial
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Peritoneal Carcinomatosis; Gastrointestinal Cancer
Keywords: cytoreductive surgery; peritoneal chemotherapy; cisplatin; cancer; gastric; biliary; pancreas; peritoneal metastases; liver metastases; peritoneal carcinomatosis from upper gastrointestinal cancer
MeSH Terms: conditions — Peritoneal Neoplasms; Gastrointestinal Neoplasms; Neoplasms | interventions — Cytoreduction Surgical Procedures; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CRS+HIPC (Experimental): Patients with biliary, gastric, or pancreatic carcinoma and metastatic or recurrent disease confined to the abdominal compartment
  Interventions: Procedure: Cytoreductive Surgery (CRS) plus Hyperthermic Intraoperative Peritoneal Chemotherapy with Cisplatin (HIPC)

INTERVENTIONS:
Procedure: Cytoreductive Surgery (CRS) plus Hyperthermic Intraoperative Peritoneal Chemotherapy with Cisplatin (HIPC) — * CRS is defined as macroscopic tumour removal using surgical resection and/or local ablative therapy (LAT)
  * HIPC is administered immediately after CRS

SUMMARY:
The majority of patients with upper gastrointestinal cancer, such as gastric, biliary, or pancreatic carcinoma, present with metastatic disease, and have an extremely poor survival, irrespective the type of treatment modality. The aim of the current monocentric phase II study is to evaluate in these patients the effectiveness of cytoreductive surgery (CRS) plus hyperthermic intraoperative peritoneal chemotherapy with cisplatin (HIPC). The study is designed to have at least 80% power to detect a 40% increase in 1-year overall survival common to all strata (gastric-biliary-pancreas) after CRS+HIPC. Over an anticipated period of 2 years, 60 patients will undergo CRS + HIPC. Translational research will quantify perioperative circulating and peritoneal tumour cells, based on real-time RT-PCR for CEA and EpCAM. Plasma concentration of cytokines will be determined for IL-1β, IL-2, IL-6, IL-8, IL-10, IL-12p70, IL-13, IFN-γ, and VEGF at several time-points. Systemic immunological changes will be assessed by flow cytometric quantification of the relative proportions and absolute numbers of B- and T-lymphocytes, NK cells, effector T cells, HLA-DR+ T cells, and regulatory T cells. Gene-expression studies will be performed using Affymetrix HG U133 Plus 2.0 arrays on primary and metastatic tissue samples.

DETAILED DESCRIPTION:
ASSESSMENT of TUMOUR BURDEN • Tumour burden will be assessed using diagnostic imaging modalities and verified by surgical or laparoscopic evaluation before CRS+HIPC

* Primary tumour Biliary adenocarcinoma

  * Intrahepatic cholangiocellular carcinoma < 3 cm in diameter
  * Extrahepatic cholangiocellular carcinoma without invasion of major blood vessels (portal vein, hepatic arteries, coeliac trunk) Gastric adenocarcinoma Macroscopic surgical margin of 5 cm is needed to obtain complete tumour removal Pancreatic adenocarcinoma Tumours located in the head, body or tail of the pancreas without portal hypertension due to complete encasement of mesenteric/portal vein and collateral venous circulation
* Liver metastases

  * Only liver metastases with stable disease or clinical response to prior systemic therapy for a period of at least 3 months are eligible
  * Not more than 3 metastases, each measuring 3 cm or less in diameter
  * Solitary liver metastasis smaller than 5 cm in diameter located in the periphery of ventral segments (Sg 2-6)
* Peritoneal metastases

  * Sugarbaker's peritoneal cancer index (PCI) will be used to assess peritoneal tumour burden 28. The completeness of cancer resection (CCR) will be assessed by the surgeon at the end of CRS; CCR-0 no macroscopic residual tumour, CCR-1 no residual tumour nodules greater than 2.5 mm, CCR-2 residual tumour nodules larger than 2.5 mm in diameter.
  * Patients with PCI < 20 are eligible for this study 11.

THERAPEUTIC INTERVENTION

* CRS is defined as macroscopic tumour removal using surgical resection and/or LAT

  o Primary tumour Biliary adenocarcinoma
* Intrahepatic cholangiocellular carcinoma

  * Deep parenchymatous tumours are treated by LAT
  * Superficial peripheral tumours are treated by resection or LAT
  * Distance between tumour and major biliary structures (right, left, main hepatic duct) needs to be > 1 cm
* Extrahepatic cholangiocellular tumours are treated by surgical resection and biliodigestive reconstruction
* Distal cholangiocellular tumours with intrapancreatic location are treated by pancreaticoduodenectomy or LAT at 90°C
* Lymph nodes around the hepatoduodenal ligament are removed Gastric adenocarcinoma
* Partial gastrectomy can be performed either by proximal or distal gastrectomy dependent on tumour location and size
* Total gastrectomy is performed in patients with signet-ring cell cancers or linitis plastica
* Tumour-draining lymph nodes are removed Pancreatic adenocarcinoma
* Tumours located in the head of the pancreas and with radiologic or macroscopic vascular invasion, which need vascular reconstruction at the time of surgery, are treated by LAT at ablation temperature of 90°C
* Tumours located in the head of the pancreas without radiologic or macroscopic vascular invasion are treated by pancreaticoduodenectomy or LAT at 90°C
* Tumours located in the body or tail of the pancreas are treated by resection or LAT of 90°C
* Tumour draining lymph nodes are removed

  o Liver metastases
* Tumours up to 3 cm are treated by LAT (RFA or MWA)
* Solitary tumour measuring 3 - 5 cm is treated by resection
* Superficial peripheral liver metastases (any diameter up to 5 cm) are allowed to be resected

  o Peritoneal metastases
* Peritonectomy, electrofulguration of superficial (< 3mm depth) metastases, and organ resection are allowed
* HIPC is administered immediately after CRS: cisplatin at a dose of 100 mg/m2 is dissolved in 3 litres of normal saline heated to less than 41° Celsius and infused into the abdominal cavity for a sustained hyperthermic intraperitoneal chemotherapy for 60 minutes. Surgical reconstruction (anastomoses) is performed after HIPC.

TRANSLATIONAL RESEARCH

1. Perioperative quantification of peritoneal and circulating tumour cells

   * Real-time qRT-PCR based on detection and quantification of CEA and EpCAM mRNA transcripts
   * Circulating tumour cells in peripheral blood samples will be studied before and at the end of surgical procedure (CRS+HIPC)
   * Peritoneal tumour cells will be evaluated in lavage fluid at the start of surgery (before any manipulation) and at the end of CRS+HIPC
2. Perioperative systemic cytokine profiles and lymphocyte immunophenotyping

   * Plasma concentration of cytokines will be determined using the BDTM Cytometric Bead Array (CBA): IL-1β, IL-2, IL-6, IL-8, IL-10, IL-12p70, IL-13, IFN-γ, and VEGF
   * The relative proportions and absolute numbers B-lymphocytes (CD19+), T-lymphocytes (CD3+), NK cells (CD56+CD3-), effector T cells (CD3+CD4+ and CD3+CD8+), HLA-DR+ T cells (CD3+HLA-DR+) and regulatory T cells (CD3+CD4+25+127low) will be quantified with flow cytometry.
   * Time-points for cytokine and immunophenotyping analyses: before surgery (d-1), at the end of surgery (d0), day after (d1) and at day 7 following CRS+HIPC
3. Gene-expression of primary and metastatic pancreatic cancer

   * To better understand cancer biology and search for novel diagnostic and therapeutic targets, fresh tissue samples from the primary tumour and from metastases will be stored in RNA-later for RNA-extraction and future analyses. Hereto, samples obtained from biliary, gastric, and pancreatic cancer tissue will be stored. Based on the fact that pancreatic cancer is associated with the worst prognosis, and based on our ongoing research on this disease, gene expression studies in the current project will be focused on pancreatic cancer.
   * In close collaboration with the department of pathology, we have stored snap-frozen tissue samples from surgically resected human pancreatic cancer for future research. Clinical, histopathological, and survival data of over 200 patients are registered in our database. Tissue samples (primary and metastases) from the current study will be analysed together with available 96 primary tumour samples that have already been controlled to be representative for high quality RNA studies. These samples are obtained from patients with early and advanced localized pancreatic cancer in various tumour stages. Gene-expression studies will be performed using Affymetrix HG U133 Plus 2.0 arrays on primary and metastatic tissue samples. These experiments will be conducted in close collaboration with the microarray facility of VIB at KUL.

ELIGIBILITY:
Inclusion Criteria:

* Primary or recurrent disease
* Histological confirmation of primary (or recurrent) and metastatic disease
* Systemic chemotherapy and/or biological is allowed before and/or after CRS+HIPC
* Radiotherapy is allowed before or after CRS+HIPC
* Patients must not have failed prior intraperitoneal platinum-therapy
* Age between 18 to 75 years
* Patient Karnofsky performance scale (KPS) > 80 (normal activity with a bit of effort)

Exclusion Criteria:

* Age < 18 or > 75 years
* Pregnancy
* Any malignancy other than biliary, gastric, or pancreatic adenocarcinoma
* Any metastatic disease outside the abdominal compartment, such as pulmonary or bone metastases
* Peritoneal carcinomatosis index (PCI) > 20 at the start of CRS
* Peritoneal residual tumour nodules larger than 2.5 mm after CRS (CCR-2)
* Clinical relevant ascites
* More than 3 liver metastases
* Solitary liver metastasis larger than 5 cm

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Overall survival time (OS) following CRS+HIPC (from surgery to cancer-related death) | 1 year follow-up
  Statistical methodology. The study is designed to have at least 80% power to detect a 40% increase in 1-y OS common to all strata (gastric-biliary-pancreas) after CRS+HIPC. The reference percentages 1-y OS are 52%, 37% and 34% for gastric, biliary and pancreatic cancer, respectively. An exponential distribution is assumed for the event times in the study group with a parameter yielding 72.8%, 51.8% and 47.6% 1-y OS in the mentioned strata.
  Cancer-specific survival will be monitored using consecutive CT- and/or MRI-scan every 3 months after CRS+HIPC.

SECONDARY OUTCOMES:
In-hospital perioperative complications | up to 24 weeks
  The number and type of perioperative complications will be recorded. The therapy-oriented severity grading system (TOSGS) of complications will be used, and complications will be allocated to surgical (SSC) and non-surgical site (NSSC) complications

CONTACTS AND LOCATIONS:
Overall Officials: Baki Topal, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Topal B, Demey K, Topal H, Jaekers J, Van Cutsem E, Vandecaveye V, Sagaert X, Prenen H. Cytoreductive surgery and Hyperthermic intra-operative peritoneal chemotherapy with Cisplatin for gastric peritoneal Carcinomatosis Monocentric phase-2 nonrandomized prospective clinical trial. BMC Cancer. 2017 Nov 17;17(1):771. doi: 10.1186/s12885-017-3730-6. PMID 29149865
- [Derived] Janky R, Binda MM, Allemeersch J, Van den Broeck A, Govaere O, Swinnen JV, Roskams T, Aerts S, Topal B. Prognostic relevance of molecular subtypes and master regulators in pancreatic ductal adenocarcinoma. BMC Cancer. 2016 Aug 12;16:632. doi: 10.1186/s12885-016-2540-6. PMID 27520560